CLINICAL TRIAL: NCT05947162
Title: Effect of Orexin System on Nicotine Addiction Among Smokers and Its Neural Mechanism
Brief Title: Effect of Orexin System on Nicotine Addiction and Its Neural Mechanism
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Kangning Hospital (Other)
Responsible Party: Principal Investigator, Huang Gengdi, Doctor, Shenzhen Kangning Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-K002-01-1
Record Dates: First submitted 2023-06-14; First posted 2023-07-17 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Tobacco Use Disorder
Keywords: nicotine; orexin; craving; withdrawal
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- smoking cessation combining with nicotine cue extinction training (Experimental): Participants should stop smoking after 18:00 the night before the test. Combined with cue exposure therapy, nicotine addicts were repeatedly presented with nicotine cue picture stimuli for extinction training, which lasted for 25 minutes.
  Interventions: Behavioral: extinction training (nicotine cues); Behavioral: Time-restricted smoking cessation
- smoking cessation combining with neutral cue extinction training (Placebo Comparator): Participants should stop smoking after 18:00 the night before the test, they are combined with cue exposure therapy, by repeatedly presenting neutral cue picture stimuli to nicotine addicts, and performing extinction training for 25 minutes.
  Interventions: Behavioral: extinction training (neutral cues); Behavioral: Time-restricted smoking cessation
- smoking cessation combining with fasting and nicotine cue extinction training (Experimental): Participants should stop smoking and eating food after 18:00 the night before the test. Combined with cue exposure therapy, nicotine addicts are repeatedly presented with nicotine cue picture stimuli for extinction training, which lasts for 25 minutes.
  Interventions: Behavioral: extinction training (nicotine cues); Behavioral: Time-restricted smoking cessation; Behavioral: Time-restricted fasting
- smoking cessation combining with fasting and neutral cue extinction training (Placebo Comparator): Participants should stop smoking and eating food after 18:00 the night before the test. Combined with cue exposure therapy, nicotine addicts were repeatedly presented with neutral cue picture stimuli for extinction training, which lasted for 25 minutes.
  Interventions: Behavioral: extinction training (neutral cues); Behavioral: Time-restricted smoking cessation; Behavioral: Time-restricted fasting
- smoking cessation combining with early lifting of fast and nicotine cue extinction training (Sham Comparator): Participants should stop smoking and eating food after 18:00 the night before the test. After breakfast at 8:00 in the morning, they are combined with cue exposure therapy, by repeatedly presenting neutral cue picture stimuli to nicotine addicts, and performing extinction training for 25 minutes.
  Interventions: Behavioral: extinction training (nicotine cues); Behavioral: Time-restricted smoking cessation; Behavioral: Time-restricted fasting with food supplemnet
- healthy control (No Intervention): Non-smoker healthy subjects matched with the smoking group in terms of age, gender, education level, etc. were used as the control group. Those healthy participants will finish fMRI scanning task.

INTERVENTIONS:
Behavioral: extinction training (nicotine cues) — extinction training: were repeatedly presented with nicotine cue picture stimuli for extinction training, which lasted for 25 minutes.
  Arms: smoking cessation combining with early lifting of fast and nicotine cue extinction training; smoking cessation combining with fasting and nicotine cue extinction training; smoking cessation combining with nicotine cue extinction training
Behavioral: extinction training (neutral cues) — extinction training: were repeatedly presented with neutral cue picture stimuli for extinction training, which lasted for 25 minutes.
  Arms: smoking cessation combining with fasting and neutral cue extinction training; smoking cessation combining with neutral cue extinction training
Behavioral: Time-restricted smoking cessation — Limiting cigarette intake within each day to a shorter interval, thus, no cigarette from 18:00 pm to 10:00 am.
  Arms: smoking cessation combining with early lifting of fast and nicotine cue extinction training; smoking cessation combining with fasting and neutral cue extinction training; smoking cessation combining with fasting and nicotine cue extinction training; smoking cessation combining with neutral cue extinction training; smoking cessation combining with nicotine cue extinction training
Behavioral: Time-restricted fasting — Limiting food intake within each day to a shorter interval, thus, no food from 18:00 pm to 10:00 am.
  Other Names: Dietary intervention
  Arms: smoking cessation combining with fasting and neutral cue extinction training; smoking cessation combining with fasting and nicotine cue extinction training
Behavioral: Time-restricted fasting with food supplemnet — Limiting food intake within each day to a shorter interval, thus, no food from 18:00 pm to 8:00 am, then supplied with breakfast.
  Other Names: Dietary intervention
  Arms: smoking cessation combining with early lifting of fast and nicotine cue extinction training

SUMMARY:
The goal of this clinical trial is to reveal the role and mechanism of orexin in nicotine addicts, compared to healthy control. The main questions it aims to answer are:

* Whether nicotine addiction-related behaviors, including nicotine withdrawal symptoms, cue-induced increased psychological craving, and relapse behavior are related to plasma orexin levels ?
* What is the neural mechanism of the orexin system in the fMRI brain network?

Participants will be asked to do as followed:

1. Day 1: Fill in the scale, test the concentration of exhaled CO, collect 5ml of blood from the vein, and take about 60 minutes.
2. Day 1-3: Test and record the amount of smoking for 3 days, about 5 minutes.
3. Day 4-5: Collect fMRI data, for about 60 minutes, perform extinction training, for about 30 minutes
4. Day 6: Fill in the scale, test the concentration of CO in exhaled breath, collect 5ml of venous blood, test after subsidence and ignition test, and collect fMRI data, for about 60 minutes.
5. Follow-up (2 weeks/4 weeks): Complete the follow-up on smoking craving and relapse by phone within 2 weeks, about 5 minutes, and complete the scale and collect fMRI data in the 4th week, about 60 minutes.

DETAILED DESCRIPTION:
Background: Smoking has always been a serious public health problem in my country. Nicotine is the main addictive ingredient in tobacco, the mechanism of nicotine addiction is not yet clear, and there is a lack of effective means to intervene in nicotine addiction. In recent years, the role of the orexin system in nicotine addiction has attracted great attention. Multiple preclinical studies have consistently found that orexin receptor antagonists have a significant intervention effect on nicotine addiction. Objective: This study focuses on the role and mechanism of orexin in nicotine addiction, and will reveal the neurobiological basis of orexin in nicotine addicts after withdrawal, and its potential as a biomarker for predicting and preventing relapse possible. Methods: This study will combine neuropsychology, neuroimaging, and detection of plasma orexin expression levels to explore whether nicotine addiction-related behaviors, including nicotine withdrawal symptoms, cue-induced increased psychological craving, and relapse behavior are related to plasma orexin Levels are associated, and further explore the neural mechanism of its brain network. Based on the detection of plasma orexin, it is of great theoretical and clinical significance to verify whether it is used as a peripheral blood biomarker of nicotine addiction and to establish an objective evaluation index of nicotine addiction. More specifically, participants need to finish following aims:

1. Scale evaluation: Minnesota Tobacco Withdrawal Symptom Scale, Smoking Craving Scale, Short Smoking Craving Questionnaire, Nicotine Dependence Level Test to evaluate nicotine dependence and Smoking Intensity Index Scale, and record the subjects' smoking index (smoking Years × number of cigarettes smoked per day/20), and the smoking craving visual analog scale was used to indicate the degree of smoking craving. In addition, the Montreal Cognitive Scale, Barratt Impulsivity Scale, Self-Rating Anxiety Scale, Self-Rating Depression Scale, Hamilton Anxiety and Depression Scale and Pittsburgh Sleep Scale were collected for about 60 minutes.
2. Behavioral extinction training: On the 4th and 5th days, combined with cue exposure therapy, nicotine addicts were repeatedly presented with nicotine cue/neutral cue picture stimulation for extinction training, which lasted for 25 minutes.
3. Collect fMRI data: including resting state fMRI and task state fMRI on the 4th and 6th day, about 60 minutes.
4. Detection of blood orexin level: 5ml of venous blood was collected on the 1st, 4th, and 6th day, and the plasma orexin-A level was measured by enzyme-linked immunosorbent assay.
5. Time and method of follow-up: Follow up the subjects through outpatient clinics, telephone, WeChat, etc., record the relapse situation within 2 weeks after the intervention, record the number of cigarettes smoked every day, and return after 1 month for nicotine withdrawal Symptoms and smoking cravings were assessed, and DTI, resting state fMRI and task state fMRI data were collected for about 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Nicotine addicts who meet the DSM-V diagnostic criteria for substance dependence, that is, smoking ≥ 10 cigarettes per day and smoking age ≥ 2 years;
2. Communicate normally with the researcher and cooperate with the researchers;

Exclusion Criteria:

1. Psychotic symptoms or a family history of mental disorders;
2. A history of dependence or behavior (gambling, online games) addiction other than alcohol, drugs, etc.;
3. Use benzodiazepines or received antipsychotic drugs within 2 weeks;
4. Epilepsy, craniocerebral injury history, coma history, brain organic or serious physical disease;
5. Body mass index (BMI) > 30 ;
6. Can not tolerate magnetic resonance examinations.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in smoking craving on Visual Analog Scale of Cigarette Craving at week 2 | baseline and week 2
  Nicotine-specific Visual Analog Scale is a valid measurements of craving for a cigarette. Possible scores range from 0 (no craving) to 10 (want cigarette imediately). Change= (Week 2 score - baseline score)
change from baseline in smoking craving on Visual Analog Scale of Cigarette Craving at week 4 | baseline and week 4
  Nicotine-specific Visual Analog Scale is a valid measurements of craving for a cigarette. Possible scores range from 0 (no craving) to 10 (want cigarette imediately). Change= (Week 2 score - baseline score)
Change from baseline in orexin level at 24 hours after administration of extinction training. | baseline and 24 hours after administration of extinction training.
  Collect 5ml of venous blood from particicpants and use a detection kit to detect orexin level.

SECONDARY OUTCOMES:
Fagerstrom Nicotine Dependence Test | baseline
  The Fagerström Test for Nicotine Dependence is a standard instrument for assessing the intensity of physical addiction to nicotine. The test was designed to provide an ordinal measure of nicotine dependence related to cigarette smoking. It contains six items that evaluate the quantity of cigarette consumption, the compulsion to use, and dependence.

CONTACTS AND LOCATIONS:
Overall Officials: Gengdi Huang, PhD, Principal Investigator — Shenzhen Kangning Hospital
Locations (1):
- Shenzhen Kangning Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No